CLINICAL TRIAL: NCT02039154
Title: The Effect of Long Duration Exercise on the Diastolic Function of the Heart
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 062012-055
Record Dates: First submitted 2013-12-10; First posted 2014-01-17 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Aging
Keywords: Exercise; Exercise tolerance; Aging; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic and strength training group (Experimental)
  Interventions: Behavioral: Aerobic and strength training group
- Balance and flexibility group (Active Comparator)
  Interventions: Behavioral: Balance and flexibility group

INTERVENTIONS:
Behavioral: Aerobic and strength training group — A exercise training program will be developed individually for each subject with the goal of increasing duration and intensity consistent with modern training techniques. Workouts will vary with respect to mode (walk, cycle, swim), duration (30-60 minutes), and intensity (base, interval, recovery) to optimize the training response. Each subject will be assigned a personal trainer and a heart rate monitor so that every session is carefully tracked and recorded. For intervals, we will use the novel high intensity aerobic intervals (HAIT). Subjects will also perform strength training 1-2 days/week.
  Arms: Aerobic and strength training group
Behavioral: Balance and flexibility group — For the balance and flexibility group, subjects will be encouraged to participate in yoga/tai chi/pilates classes that is approved by one of the exercise physiologists on the research team. The goal for this group is exercise classes that will be of benefit to them, but that will not include sustained aerobic, endurance exercise. In place of a group exercise class, subjects will have the option of purchasing videos for home use. The subjects will be encouraged to participate in some form of non-endurance training at least 3 days per week. Each subject will receive an exercise log in which they will be expected to record their training.
  Arms: Balance and flexibility group

SUMMARY:
The purpose of this study is to determine whether vigorous exercise training 4-5 days/week for 2 years in sedentary middle aged men and women (ages 45-64) will improve cardiac and vascular compliance to a degree equivalent to life-long exercisers and the sedentary young. Sedentary aging is associated with impaired diastolic function, which can lead to heart failure. However, if exercise training can be implemented early enough in life while cardiovascular plasticity still exists, then functional capacity can be maintained, preventing heart failure.

DETAILED DESCRIPTION:
Objectives: Chronic physical inactivity contributes to the deaths of nearly 1 in 10 Americans. In seniors, the single most common life-threatening disease is congestive heart failure and for these patients, abnormalities of diastolic function play a critical role in the pathophysiology of their disease. The primary investigator's previous research has demonstrated that: a) healthy but sedentary aging leads to atrophy and stiffening of the heart with reduced myocardial and chamber compliance; b) in contrast, highly competitive senior athletes had cardiac compliance that was indistinguishable from healthy young individuals suggesting that lifelong exercise training prevented this stiffening; c) even prolonged and intense exercise training started after age 65 failed to reverse age-related cardiac and vascular stiffening; d) cardiac stiffening begins in middle age (45-64) and can be substantially prevented by training 4-5 days/wk. The primary objective of this project, is therefore to identify sedentary individuals aged 45-64, and initiate an exercise program carefully designed to maximize effects on cardiovascular compliance and function. After this aim is accomplished, we will have established a novel, practical exercise training strategy designed to prevent the cardiovascular stiffening with aging, improve the functional capacity in our aging population, and ultimately to prevent Heart failure with preserved Ejection Fraction. Such a determination would have enormous public health significance since this condition is quite difficult to treat once established.

Hypothesis: The investigators hypothesize that exercise training implemented 4-5 times/week for 2 yrs in sedentary middle aged men and women (45-64yr) will improve cardiac and vascular compliance to a degree equivalent to life-long exercisers (and sedentary young). The investigators will perform invasive and non-invasive assessment of cardiovascular structure and function before and after an exercise program involving high intensity aerobic intervals, lower intensity endurance ("base training"), and strength training.

Specific Aim: To test our hypothesis, there will be two groups of previously sedentary subjects, ages 45-64 for 2 years, with the following interventions: 1) subjects undergoing prolonged endurance/interval/strength exercise training; and 2) yoga/balance control.

A comprehensive set of "Baseline Testing" (prior to the two year intervention) and "Follow-up Testing" (after the two year intervention) will take place to assess the effects of the intervention. This testing will include submaximal and maximal exercise testing as well as comprehensive invasive (right heart catheterization) and non-invasive (ultrasound) measures of cardiac mechanics, relaxation and morphology. From these data, the following indices of diastolic and systolic function will be generated: Starling and pressure/volume curves; calculations of left ventricle wall stress and strain; and measurements of flow propagation velocity, ejection fraction and relaxation velocity.

ELIGIBILITY:
Inclusion Criteria:

* healthy, sedentary men and women
* ages 45-64
* body mass index <30
* absence of co-morbid conditions including hypertension, diabetes, heart failure, asthma, chronic obstructive pulmonary disease, coronary artery disease as evidenced by angina or prior myocardial infarction or cerebrovascular disease as evidenced by prior transient ischemic attack or stroke

Exclusion Criteria:

* healthy, active (aerobic exercisers greater than 2 days per week) men and women
* ages less than 45 or over 64
* body mass index >30
* presence of co-morbid conditions including hypertension, diabetes, heart failure, asthma, chronic obstructive pulmonary disease, coronary artery disease as evidenced by angina or prior myocardial infarction or cerebrovascular disease as evidenced by prior transient ischemic attack or stroke
* Patients with chronic orthopedic injury that might make them unable to participate in an exercise testing will also be excluded
* Subjects unable to speak English will not be recruited because of the complex experimental studies and the need for precise communication between the volunteers and the research staff to ensure safety.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular stiffness (diastolic function/static) after training | Two years

SECONDARY OUTCOMES:
Change in diastolic function/dynamic after training | 2 years
Change in systolic function after training | 2 years
Change in ventricular-vascular coupling after training | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

REFERENCES:
- [Derived] Hieda M, Sarma S, Hearon CM Jr, Dias KA, Martinez J, Samels M, Everding B, Palmer D, Livingston S, Morris M, Howden E, Levine BD. Increased Myocardial Stiffness in Patients With High-Risk Left Ventricular Hypertrophy: The Hallmark of Stage-B Heart Failure With Preserved Ejection Fraction. Circulation. 2020 Jan 14;141(2):115-123. doi: 10.1161/CIRCULATIONAHA.119.040332. Epub 2019 Dec 23. PMID 31865771
- [Derived] McNamara DA, Aiad N, Howden E, Hieda M, Link MS, Palmer D, Samels M, Everding B, Ng J, Adams-Huet B, Opondo M, Sarma S, Levine BD. Left Atrial Electromechanical Remodeling Following 2 Years of High-Intensity Exercise Training in Sedentary Middle-Aged Adults. Circulation. 2019 Mar 19;139(12):1507-1516. doi: 10.1161/CIRCULATIONAHA.118.037615. PMID 30586729
- [Derived] Opondo MA, Aiad N, Cain MA, Sarma S, Howden E, Stoller DA, Ng J, van Rijckevorsel P, Hieda M, Tarumi T, Palmer MD, Levine BD. Does High-Intensity Endurance Training Increase the Risk of Atrial Fibrillation? A Longitudinal Study of Left Atrial Structure and Function. Circ Arrhythm Electrophysiol. 2018 May;11(5):e005598. doi: 10.1161/CIRCEP.117.005598. PMID 29748195
- [Derived] Howden EJ, Sarma S, Lawley JS, Opondo M, Cornwell W, Stoller D, Urey MA, Adams-Huet B, Levine BD. Reversing the Cardiac Effects of Sedentary Aging in Middle Age-A Randomized Controlled Trial: Implications For Heart Failure Prevention. Circulation. 2018 Apr 10;137(15):1549-1560. doi: 10.1161/CIRCULATIONAHA.117.030617. Epub 2018 Jan 8. PMID 29311053